CLINICAL TRIAL: NCT00954343
Title: Shockwave Treatment of Diabetic Foot Ulcer. A Prospective, Controlled, Randomized Trial. Step 1
Brief Title: Shockwave Treatment of Diabetic Foot Ulcer: Step I
Acronym: STUF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2456/09
Record Dates: First submitted 2009-07-31; First posted 2009-08-07 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Diabetic Foot Ulcers
Keywords: Foot Ulcers; Extracorporeal Shockwave; Chronic wound
MeSH Terms: conditions — Foot Ulcer | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group I (Experimental)
  Interventions: Procedure: Extracorporeal Shock Wave
- Group II (Experimental)
  Interventions: Procedure: Extracorporeal Shock Wave
- Group III (Experimental)
  Interventions: Procedure: Extracorporeal Shock Wave
- Group IV (Experimental)
  Interventions: Procedure: Extracorporeal Shock Wave
- Group V (No Intervention)

INTERVENTIONS:
Procedure: Extracorporeal Shock Wave
  Arms: Group I
Procedure: Extracorporeal Shock Wave
  Arms: Group II
Procedure: Extracorporeal Shock Wave
  Arms: Group III
Procedure: Extracorporeal Shock Wave
  Arms: Group IV

SUMMARY:
Extracorporeal Shock Wave treatment is a well established treatment in orthopedics. Considerable success has been reported after treatment of various soft tissue pathologies (Tendinitis, heel spur etc). In recent years, encouraging results have been reported concerning the effect of the shock-wave on chronic wounds. It has been reported that healing time can be considerably shortened if shock-waves are applied to the wound in addition to conventional wound treatment. Yet, randomized, controlled, prospective trials are missing.

In this study, the effect of shock-waves on diabetic foot ulcer shall be assessed.

The study is composed of 5 groups of which 4 groups receive shock wave treatments (each with a different protocol). One group serves as an untreated control group. All groups get standardized wound treatment and wound dressing.

That shock-wave application protocol that shows the best results (rate of completely healed ulcer, most decrease of ulcer size) shall be tested in a further, sufficiently dimensioned, two-armed, randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Diabetes Type I or II
* Chronic ulcer on the foot
* Ulcer present for at least 6 weeks
* Wagner Grade 1 or 2

Exclusion Criteria:

* Chronic rest pain
* Critical ischemia
* Gangrene
* Ankle-Arm-Index < 0,5
* Critical ischemia treated within 6 weeks before possible enrollment
* Ulcer of Grade 3 or worse according to the Wagner Classification
* Osteomyelitis
* Affection of toes
* Necessity of surgical intervention
* Malalignment of the foot sustaining the ulcer
* Treatment of Ulcer with Prostaglandins or vasodilatators within the last 2 weeks
* Current therapy with corticoids
* Infection with HIV; Hepatitis
* Suppression of immune system (due to illness or medication)
* Medication with Vitamin-K-Antagonists
* Known hemophilia
* Sever Hypalbuminemia < 2 g/dl
* Severe anemia
* Ulcer other than of diabetic origin
* Pregnant or breast-feeding women
* Known coagulopathies
* Implants such as artificial heart valves, joint replacement, bone replacement, osteosynthesis material
* Patients participating on other studies
* Chemotherapy within the last 60 days
* Mentally disabled patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08

PRIMARY OUTCOMES:
Percentage decrease of ulcer size twelve weeks after treatment begin (i.e. first shock wave treatment) compared to the baseline (ulcer size at first treatment)

SECONDARY OUTCOMES:
Rate of completely healed ulcer 6, 9 and 12 weeks after first treatment
Percentage decrease of ulcer size 6 and 9 weeks after first treatment
Tissue oxygen concentration after shock wave treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gollwitzer, PD Dr., CCRP, Principal Investigator — Klinik für Orthopädie und Unfallchirurgie Klinikum rechts der Isar
Locations (1):
- Klinik für Orthopädie und Unfallchirurgie, Klinikum rechts der Isar, Munich, Bavaria, Germany